CLINICAL TRIAL: NCT01481909
Title: Study on Mastocytosis for Rupatadine Treatment An Exploratory Phase IV, Randomised, Double-blind, Placebo Controlled Crossover Study to Assess the Efficacy of 20 mg Rupatadine on the Treatment of
Brief Title: Study on Mastocytosis for Rupatadine Treatment
Acronym: SMART
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Marcus Maurer (Other)
Responsible Party: Sponsor-Investigator, Marcus Maurer, Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMART-2010-1
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Mastocytosis
Keywords: Assessment of wheal and flare development; Assessment of life quality
MeSH Terms: conditions — Mastocytosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): All patients included in this study will be subjected at the screening visit to a standardized provocation of Darier's sign by a device for standardized provocation testing (Hartmann and Siebenhaar 2009). Patients that exhibit positive skin test reactions will be enrolled, provided that they meet all inclusion criteria and none of the exclusion criteria and that they give informed consent. Study patients will receive treatment for 28 days (minimal 25, maximal 30 days) before visit 1 and visit 2 including the same day before the provocation test (RUP 20mg/day or placebo according to randomization). All patients will receive antihistaminic rescue medication immediately after completing the testing when necessary.
  Interventions: Drug: Rupatadin
- Rupafin (Active Comparator): All patients included in this study will be subjected at the screening visit to a standardized provocation of Darier's sign by a device for standardized provocation testing (Hartmann and Siebenhaar 2009). Patients that exhibit positive skin test reactions will be enrolled, provided that they meet all inclusion criteria and none of the exclusion criteria and that they give informed consent. Study patients will receive treatment for 28 days (minimal 25, maximal 30 days) before visit 1 and visit 2 including the same day before the provocation test (RUP 20mg/day or placebo according to randomization). All patients will receive antihistaminic rescue medication immediately after completing the testing when necessary.
  Interventions: Drug: Rupatadin

INTERVENTIONS:
Drug: Rupatadin — 20 mg, 28 days over 60 days
  Other Names: Each tablet contains 10 mg RUP

SUMMARY:
Study title:

An exploratory, randomised, double-blind, placebo controlled crossover study to assess the efficacy of 20 mg Rupatadine on the treatment of mastocytosis symptoms.

Study code:

SMART-2010-1 Principal Investigator, Co-Investigator, sponsor, and study centre (acc. to § 40 Abs. 4 AMG) Dr. med. F. Siebenhaar, Prof. Dr. Med. M. Maurer, Allergie-Centrum-Charité, Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin, Charitéplatz 1, D-10117 Berlin Biometry and biostatistical analyses Division of Biostatistics and Clinical Epidemiology, Charité - Universitätsmedizin Berlin, Charitéplatz 1, D-10117 Berlin Monitoring Coordination Centre for Clinical Studies (KKS), Charité - Universitätsmedizin Berlin, Charitéplatz 1, D-10117 Berlin Clinical phase Phase II

Primary objective:

Reduction of wheal and flare type skin reaction after standardised provocation testing assessed by volumetric and thermographic measurements.

Secondary objectives:

Improvement of additional related symptoms (e.g. pruritus) and subjective affliction as assessed by symptom score, DLQI, Itchy-QoL and VAS.

Study design:

An exploratory, randomised, double-blind, placebo controlled crossover study

Type and number of patients:

Male and female patients (n = 30) with cutaneous mastocytosis and indolent systemic mastocytosis with skin involvement

Main criteria for inclusion:

Mastocytosis patients aged 18-65 years, signed written consent, no systemic corticosteroid or other immunosuppressive therapy, no permanent severe diseases Test product, dose and mode of administration 20 mg Rupatadine or placebo before provocation testing, oral administration (tablets)

Duration of treatment:

28 days (testing will be done at the day of last treatment)

Assessment of efficacy:

1. Assessment of wheal and flare development by planimetric analyses of digital photographic, volumetric, and thermographic imaging (time lapse) before and after treatment with study medication,
2. Additional assessment of symptoms,
3. Assessment of life quality

Main criteria of evaluation:

Efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stable symptomatic maculopapulous cutaneous mastocytosis or indolent systemic mastocytosis with skin involvement and a positive Darier's Sign
2. Age between 18 and 65 years.
3. Female patients must be using a highly effective method of birth control (such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence, vasectomised partner), or they must be postmenopausal, surgically sterilised, or hysterectomised.
4. Voluntarily signed written informed consent.

Exclusion Criteria:

1. The presence of permanent severe diseases, especially those affecting the immune system, except for mastocytosis
2. History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
3. History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy, hyper-/hypokalemia, bradycardia < 50bpm, QTc interval > 440ms
4. Evidence of severe renal dysfunction (creatinine > 1,5 x upper reference value)
5. Evidence of significant hepatic disease (liver enzymes > 2 x upper reference value)
6. History of adverse reactions to RUP, or other ingredients of the IMP
7. Presence of active cancer which requires chemotherapy or radiation therapy
8. Aggressive systemic mastocytosis
9. History or presence of alcohol abuse or drug addiction
10. Participation in any clinical trial within 4 weeks prior to enrolment
11. Commitment to an institution in terms of § 40 Abs. 1 S. 3 Nr. 4 AMG
12. Intake of antihistamines or leukotriene antagonists within 7 days prior to the beginning of the study
13. Intake of oral corticosteroids within 14 days prior to the beginning of the study
14. Use of depot corticosteroids or chronic systemic corticosteroids within 21 days before beginning of the study
15. Pregnancy or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pruritus | 10 weeks
  Reduction of pruritus and wheal and flare type skin reaction after standardised provocation testing as assessed by volumetric and thermographic measurements.

SECONDARY OUTCOMES:
Questionaire | 10 weeks
  Improvement of additional disease related symptoms and subjective affliction as measured by physician and patient global assessments, DLQI, Itchy-QoL and QoL(i)MaP*.
  *not validated questionnaire for mastocytosis symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — University Berlin Charitè
Locations (1):
- University Charité, Berlin, Germany, Germany